CLINICAL TRIAL: NCT00825357
Title: Biological Markers to Identify Early Sepsis and Acute Lung Injury
Status: Completed | Type: Observational
Sponsor: Chimei Medical Center (Other)
Responsible Party: Principal Investigator, Kuo-Chen Cheng, Chief, Chimei Medical Center
Other Study IDs: CM-IRB09509002
Record Dates: First submitted 2009-01-15; First posted 2009-01-21 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Sepsis; Acute Lung Injury
Keywords: biological markers; sepsis; acute lung injury
MeSH Terms: conditions — Sepsis; Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There are no clear markers to identify sepsis and acute lung injury at early stage in clinical settings which would result in improved survival of the patients. In collaboration with the research team led by Dr. Zhang at St. Michael's Hospital, Toronto, we have initiated a pilot study looking for biological markers to detect severe sepsis and ARDS. We have found that human neutrophils peptides (a-defensins), certain coagulation variables and cytokine levels are very sensitive markers to differentiate severe sepsis, ARDS from cardiovascular diseases in ICU patients. These findings may provide valuable information for therapeutic guideline in clinical practice. The present study will focus on testing 'biological markers' to identify patients with sepsis and acute lung injury. We will examine the roles of three components of markers including inflammation, neutrophil activation and coagulation. We are hoping that this proposed translational research will help develop novel therapeutic strategy in sepsis and acute lung injury patients.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria of ≧2 SIRS or acute lung injury.
* Get agreement of patient's attending physician and inform consent form patient or family.

Exclusion Criteria:

* Use Antibiotics over 24 hrs（only SIRS group）.
* Active bleeding.
* Pregnancy.
* Active Cancer (refer to malignancy which is recently diagnosed, under treatment, or relapsed)
* VS or Subject or Family refuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU and age ≧18-year-old.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The present study will focus on testing 'biological markers' to identify patients with sepsis and acute lung injury in early stage. | 72 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Intensive Care Medicine; Chi Mei Medical Center, Tainan, Taiwan